CLINICAL TRIAL: NCT01920893
Title: A Randomized, Double-Blind, Phase 2, Placebo Controlled, 2 Arm Study To Evaluate Dupilumab In Patients With Bilateral Nasal Polyposis And Chronic Symptoms Of Sinusitis
Brief Title: An Evaluation of Dupilumab in Patients With Nasal Polyposis And Chronic Symptoms Of Sinusitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT12340; 2013-001803-35 (EudraCT Number); U1111-1130-6475 (Other: UTN)
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — dupilumab; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for dupilumab), 2 subcutaneous injections on Day 1 as a loading dose followed by a single injection every week (QW) from Week 1 to 15 added to Mometasone furoate nasal spray (MFNS).
  Interventions: Drug: Placebo (for dupilumab); Drug: Mometasone furoate nasal spray
- Dupilumab 300 mg QW (Experimental): Dupilumab, 2 Subcutaneous injections on Day 1 as a loading dose for a total of 600 mg, followed by a single 300 mg injection QW from Week 1 to 15 added to MFNS.
  Interventions: Drug: Dupilumab; Drug: Mometasone furoate nasal spray

INTERVENTIONS:
Drug: Placebo (for dupilumab) — Solution for injection; Subcutaneous injection.
  Arms: Placebo
Drug: Dupilumab — Solution for injection; Subcutaneous injection.
  Other Names: SAR231893; REGN668
  Arms: Dupilumab 300 mg QW
Drug: Mometasone furoate nasal spray — Nasal spray, 2 actuations in each nostril twice daily.
  Other Names: NASONEX®

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab (SAR231893/REGN668) in the treatment of bilateral Nasal Polyposis (NP) by assessment of the endoscopic nasal polyp score (NPS) in comparison to placebo.

Secondary Objectives:

To evaluate effect of dupilumab with regards to:

* symptoms of sinusitis,
* sinus computed tomography (CT) scan,
* NPS in the sub-group of participants with co-morbid asthma,
* Safety and tolerability.

DETAILED DESCRIPTION:
Screening period (4 weeks) + Randomized Treatment Period (16 weeks) + Post-Treatment Period (16 weeks) = 36 weeks.

To ensure at least 28 participants with co-morbid asthma needed for subgroup analysis, recruitment of NP participants without co-morbid asthma would stop when approximately 28 participants without asthma were randomized.

ELIGIBILITY:
Inclusion criteria: participants with:

* A minimum bilateral nasal polyp score of 5 out of a maximum score of 8 (with a unilateral score of at least 2 for each nostril) despite completion of a prior intranasal corticosteroid (INCS) treatment for at least 8 weeks before screening.
* Presence of at least two of the following symptoms prior to screening: nasal blockade/obstruction/congestion or nasal discharge (anterior/posterior nasal drip); facial pain/pressure; reduction or loss of smell.

Exclusion criteria:

* Participants <18 or >65 years of age.
* Sinonasal outcome test (SNOT-22) <7.
* Participants who had taken other investigational drugs or prohibited therapy for this study within 2 months before screening or 5 half-lives, whichever was longer:

  * Burst of systemic corticosteroids within the 2 months before screening or were scheduled to receive systemic corticosteroids during the study period for another condition
  * INCS drops within 1 month prior to screening
  * Monoclonal antibody (mAB) and immunosuppressive treatment
  * Anti-immunoglobulin E (IgE) therapy (omalizumab) within 130 days of Visit 1
  * Leukotriene antagonists/modifiers unless participant was on a continuous treatment for at least 30 days prior to Visit 1.
* Participants who had undergone any nasal surgery (including polypectomy) within 6 months before screening or have had more than 5 sinonasal surgeries in the past of which maximal 2 were surgeries changing the lateral wall structure of the nose.
* Participants with asthma having:

  * Forced Expiratory Volume (FEV1) ≤ 60%, or .Asthma exacerbation requiring systemic (oral and/or parenteral) steroid treatment or hospitalization for >24 hours for treatment of asthma, within 3 months prior to screening or were on a dose of greater than 1000 microgram (mcg) fluticasone or an equivalent INCS.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- United States (5):
  - Investigational Site Number 840014, Rolling Hills Estates, California
  - Investigational Site Number 840015, Denver, Colorado
  - Investigational Site Number 840013, Boston, Massachusetts
  - Investigational Site Number 840002, Lake Oswego, Oregon
  - Investigational Site Number 840009, Pittsburgh, Pennsylvania
- Belgium (2):
  - Investigational Site Number 056001, Ghent
  - Investigational Site Number 056002, Leuven
- Spain (5):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724003, Faitanar
  - Investigational Site Number 724005, Jerez de la Frontera
  - Investigational Site Number 724002, L'Hospitalet de Llobregat
  - Investigational Site Number 724004, Madrid
- Sweden (2):
  - Investigational Site Number 752001, Stockholm
  - Investigational Site Number 752002, Stockholm

REFERENCES:
- [Result] Bachert C, Mannent L, Naclerio RM, Mullol J, Ferguson BJ, Gevaert P, Hellings P, Jiao L, Wang L, Evans RR, Pirozzi G, Graham NM, Swanson B, Hamilton JD, Radin A, Gandhi NA, Stahl N, Yancopoulos GD, Sutherland ER. Effect of Subcutaneous Dupilumab on Nasal Polyp Burden in Patients With Chronic Sinusitis and Nasal Polyposis: A Randomized Clinical Trial. JAMA. 2016 Feb 2;315(5):469-79. doi: 10.1001/jama.2015.19330. PMID 26836729
- [Derived] Khan AH, Abbe A, Falissard B, Carita P, Bachert C, Mullol J, Reaney M, Chao J, Mannent LP, Amin N, Mahajan P, Pirozzi G, Eckert L. Data Mining of Free-Text Responses: An Innovative Approach to Analyzing Patient Perspectives on Treatment for Chronic Rhinosinusitis with Nasal Polyps in a Phase IIa Proof-of-Concept Study for Dupilumab. Patient Prefer Adherence. 2021 Nov 19;15:2577-2586. doi: 10.2147/PPA.S320242. eCollection 2021. PMID 34848949
- [Derived] Khan AH, Reaney M, Guillemin I, Nelson L, Qin S, Kamat S, Mannent L, Amin N, Whalley D, Hopkins C. Development of Sinonasal Outcome Test (SNOT-22) Domains in Chronic Rhinosinusitis With Nasal Polyps. Laryngoscope. 2022 May;132(5):933-941. doi: 10.1002/lary.29766. Epub 2021 Aug 26. PMID 34437720
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614
- [Derived] Boyle JV, Lam K, Han JK. Dupilumab in the treatment of chronic rhinosinusitis with nasal polyposis. Immunotherapy. 2020 Feb;12(2):111-121. doi: 10.2217/imt-2019-0191. Epub 2020 Feb 20. PMID 32075470
- [Derived] Bachert C, Hellings PW, Mullol J, Hamilos DL, Gevaert P, Naclerio RM, Joish VN, Chao J, Mannent LP, Amin N, Abbe A, Taniou C, Fan C, Pirozzi G, Graham NMH, Mahajan P, Staudinger H, Khan A. Dupilumab improves health-related quality of life in patients with chronic rhinosinusitis with nasal polyposis. Allergy. 2020 Jan;75(1):148-157. doi: 10.1111/all.13984. Epub 2019 Oct 23. PMID 31306495
- [Derived] Laidlaw TM, Mullol J, Fan C, Zhang D, Amin N, Khan A, Chao J, Mannent LP. Dupilumab improves nasal polyp burden and asthma control in patients with CRSwNP and AERD. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2462-2465.e1. doi: 10.1016/j.jaip.2019.03.044. Epub 2019 Apr 4. No abstract available. PMID 30954643
- [Derived] Jonstam K, Swanson BN, Mannent LP, Cardell LO, Tian N, Wang Y, Zhang D, Fan C, Holtappels G, Hamilton JD, Grabher A, Graham NMH, Pirozzi G, Bachert C. Dupilumab reduces local type 2 pro-inflammatory biomarkers in chronic rhinosinusitis with nasal polyposis. Allergy. 2019 Apr;74(4):743-752. doi: 10.1111/all.13685. Epub 2019 Jan 21. PMID 30488542

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 sites in 4 countries. A total of 60 participants were randomized between August 2013 and March 2014.
Pre-assignment Details: Randomization was stratified according to medical history of asthma (with/without asthma) and by nasal biopsy (biopsy performed,Yes/No). Assignment was done centrally using Interactive Voice/Web Response System in 1:1 ratio (dupilumab:placebo)after 4-week run-in period on Mometasone furoate nasal spray (MFNS) and confirmation of selection criteria.
Groups:
- Placebo: Placebo (for dupilumab), 2 subcutaneous injections on Day 1 as a loading dose followed by a single injection every week (QW) from Week 1 to 15 added to MFNS.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg QW
Started | 30 | 30
Treated (Safety Population) | 30 | 30
Completed | 23 | 28
Not Completed | 7 | 2
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Placebo: Placebo (for dupilumab), 2 subcutaneous injections on Day 1 as a loading dose followed by a single injection QW from Week 1 to 15 added to MFNS.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg QW | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (9.1) | 47.4 (9.8) | 48.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 16 | 18 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 30 | 28 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Number of participants with asthma [Count of Participants; unit: Participants] — The diagnosis of asthma was based on participant's history; participants with asthma were required to have a forced expiratory volume in 1 second (FEV1) of more than 60% of predicted use, daily inhaled corticosteroids of no more than 1000 mcg of fluticasone (or equivalent), and could not have had an asthma exacerbation requiring systemic corticosteroids or hospitalization within the prior 3 months.
  Participants
    Yes | 19 | 16 | 35
    No | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bilateral Endoscopic Nasal Polyp Score (NPS) at Week 16
Description: NPS was the sum of the right and left nostril scores, as evaluated by means of nasal endoscopy. Total score ranges from 0 to 8 (scored 0 [no polyp] to 4 [large polyps] for each nostril), with a lower score indicating smaller-sized polyps.
Time Frame: Baseline, Week 16
Population: Intent-to-treat (ITT) population included all randomized participants analyzed according to the treatment group allocated by randomization. Here, number analyzed = number of participants with available data for specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 5.67 (0.88) | 5.87 (1.01)
  Week 16: number analyzed (Participants) | 23 | 29
  Week 16 | 5.39 (1.47) | 3.97 (1.9)
  Change from baseline at Week 16: number analyzed (Participants) | 23 | 29
  Change from baseline at Week 16 | -0.26 (1.32) | -1.9 (1.76)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab 300 mg QW; Analysis was performed by a mixed model repeated measures (MMRM) model; Test type: Superiority; p = 0.0009, Mixed Models Analysis — Threshold for significance at 0.05 level; Least Square (LS) mean difference = -1.55, 95% CI 2-sided [-2.43 to -0.67] — Dupilumab 300 mg QW vs Placebo

2. Secondary Outcome: Change From Baseline in Bilateral Endoscopic NPS at Week 16 in Participants With Asthma
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: Participants of the ITT population with asthma and with available data at Week 16.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 15 | 15
score on a scale | 0.27 (0.88) | -2.4 (2.03)

3. Secondary Outcome: Change From Baseline in Participant Reported Symptoms Scores of Sinusitis at Week 16
Description: Morning symptoms of sinusitis (nasal congestion/obstruction, anterior rhinorrhea [runny nose], posterior rhinorrhea [post nasal drip], and loss of sense of smell) were assessed using a 0 (no symptoms) - 3 (severe symptoms) categorical scale where higher score indicated severe symptoms.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with data available for symptom score at Week 16.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 23 | 29
score on a scale
  Congestion/obstruction | -0.26 (0.7) | -0.95 (0.86)
  Runny nose | -0.1 (0.58) | -0.62 (0.9)
  Post nasal drip | -0.15 (0.59) | -0.49 (0.78)
  Loss of sense of smell | -0.3 (0.6) | -1.36 (1.08)

4. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) for Rhinosinusitis Symptoms Severity at Week 16
Description: Severity of rhinosinusitis symptoms were assessed on a 0 cm (not troublesome) - 10 cm (worst thinkable troublesome) VAS where higher score indicated worst thinkable troublesome.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with data available for Rhinosinusitis Symptoms Severity VAS at Week 16.
Measure: Mean (Standard Deviation); unit: centimetre (cm)
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 19 | 28
centimetre (cm) | -1.84 (3.6) | -4.32 (2.75)

5. Secondary Outcome: Change From Baseline in Nasal Peak Inspiratory Flow (NPIF) at Week 16
Description: NPIF evaluation represents a physiologic measure of the air flow through both nasal cavities during forced inspiration and/or expiration expressed in liter per minute.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with data available for NPIF at Week 16.
Measure: Mean (Standard Deviation); unit: liter/minute
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 23 | 29
liter/minute
  NPIF-Morning | 28.81 (34.26) | 61.91 (43.39)
  NPIF-Evening | 26.65 (34.31) | 61.25 (45.91)

6. Secondary Outcome: Change From Baseline in Smell Test (University of Pennsylvania Smell Identification Test [UPSIT]) Scores at Week 16
Description: UPSIT was a 40-item test to measure the individual's ability to detect odors. Total score ranges from 0 (anosmia)-40 (normal sense of smell), lower score indicated severe smell loss.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with data available for UPSIT at Week 16.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 23 | 28
score on scale | -0.17 (5.1) | 15.36 (9.61)

7. Secondary Outcome: Change From Baseline in Sinus Computed Tomography (CT) Scan Assessments at Week 16: Lund-Mackay Score
Description: CT scan assessment included Lund-Mackay score and percent of the maxillary sinuses occupied by disease. The Lund-Mackay scoring system rated each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses. The total score ranges from 0 (normal) - 24 (more opacified); higher score indicated worse status.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with CT scan data available at Week 16.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 26 | 29
score on scale | -0.23 (3.74) | -9.24 (4.58)

8. Secondary Outcome: Change From Baseline in Sinus Computed Tomography (CT) Scan Assessments at Week 16: Percent Area Occupied by Disease
Description: CT scan assessment included Lund-Mackay score and percentage of the area of maxillary sinuses occupied by disease.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with CT scan data available at Week 16.
Measure: Mean (Standard Deviation); unit: percent area
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 26 | 29
percent area | -3.92 (20.54) | -35.66 (24.28)

9. Secondary Outcome: Time to First Response in NPS: Kaplan-Meier Estimate at Week 16
Description: The time-to-first response in NPS: time from the date of randomization to the date of first NPS (defined as >=1 point reduction from baseline score); for participants without NPS >=1 point reduction, it was censored at the end of treatment date. The median time to first response was not estimated because the number of responses was too low in the Dupilumab arm. Therefore, alternative Kaplan-Meier statistics, the probability of response at Week 16, are presented as the descriptive measure statistics.
Time Frame: Baseline to Week 16
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Probability of response
Groups:
- Dupilumab 300 mg QW: Dupilumab, 2 subcutaneous injections on Day 1 as a loading dose for a total of 600 mg, followed by a single 300 mg injection every week from Week 1 to 15 added to MFNS.
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 30
Probability of response | 0.44 [0.242 to 0.638] | 0.828 [0.69 to 0.965]

10. Secondary Outcome: Change From Baseline in 22-Item Sinonasal Outcome Test (SNOT-22) at Week 16
Description: The SNOT-22 was a validated questionnaire to assess the impact of chronic rhinosinusitis on quality of life. The total score may range from 0 (no problem)-110 (worst quality of life), higher scores represented worst quality of life; minimal clinically important change ≥ 8.90.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with SNOT-22 data available at Week 16.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 23 | 29
score on a scale | -8.26 (17.63) | -29.1 (19.9)

11. Post Hoc Outcome: Change From Baseline in Nasal Total Symptoms Score (nTSS) at Week 16
Description: nTSS was the sum of participant-assessed nasal symptom scores for nasal congestion/obstruction, decreased/loss of sense of smell, and rhinorrhea (anterior/posterior nasal discharge), each accessed on 0-3 categorical scale. Total score ranges from 0 (no symptoms) to 9 (severe symptoms). Higher score indicated severe symptoms.
Time Frame: Baseline, Week 16
Population: Participants from ITT population with nTSS data available at Week 16.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Dupilumab 300 mg QW
Number analyzed (Participants) | 23 | 29
score on a scale
  nTSS - Morning | -0.68 (1.44) | -2.87 (2.09)
  nTSS - Evening | -0.77 (1.48) | -2.9 (2.04)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 32) regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: Reported AEs and deaths are treatment emergent AEs that developed/worsened and deaths that occurred during the 'treatment emergent period' (from the first dose of the double-blind IMP injection up to the end of the 16 weeks post-treatment period).
Groups:
- Placebo: Participants exposed to placebo (for dupilumab) added to MFNS (mean exposure of 14 weeks).
- Dupilumab 300 mg QW: Participants exposed to dupilumab added to MFNS (mean exposure of 16 weeks).
Arm/Group | Placebo | Dupilumab 300 mg QW
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30 | 2/30
Other Adverse Events (participants affected / at risk) | 22/30 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Dupilumab 300 mg QW (N=30)
Herpes zoster (Infections and infestations) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Dupilumab 300 mg QW (N=30)
Bronchitis (Infections and infestations) | 4 | 1
Nasopharyngitis (Infections and infestations) | 10 | 14
Sinusitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 5 | 6
Sinus headache (Nervous system disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Injection site reaction (General disorders) | 2 | 12
Blood creatine phosphokinase increased (Investigations) | 2 | 0

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of participants analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.